CLINICAL TRIAL: NCT06621979
Title: Evaluation of Post-Omega Bypass Excluded Stomach Fundoplication to Treat Disabling Gastroesophageal Reflux Disease Resistant to Medical Treatment and Requiring Surgery
Brief Title: Evaluation of the Fundoplicature of the Excluded Stomach Post Omega Bypass
Acronym: FEE-RGOIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A02501-44
Record Dates: First submitted 2024-09-30; First posted 2024-10-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Bypass, Gastric

STUDY DESIGN:
Intervention Model Description: Single-center, ambispective, interventional, non-randomized pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastroesophageal reflux disease (Experimental): Disabling post-bypass gastroesophageal reflux, resistant to medical treatment and requiring surgery
  Interventions: Procedure: Bypass surgery type one anastomosis gastric bypass

INTERVENTIONS:
Procedure: Bypass surgery type one anastomosis gastric bypass — Adult patients who have undergone single-anastomosis gastric bypass followed by fundoplication of the excluded stomach for the treatment of disabling post-bypass gastroesophageal reflux, resistant to medical treatment and requiring surgical intervention.

SUMMARY:
The purpose of this study is to evaluate the efficacy of fundoplication with stomach excluded in the suppression of disabling gastroesophageal reflux requiring surgery in patients who have undergone one anastomosis gastric bypass, with complete objective evaluation of reflux.

DETAILED DESCRIPTION:
The FEE& RGOIC trial is a single-center, ambispective, interventional, non-randomized pilot study to evaluate the efficacy of Fundoplicature with stomach excluded objectively and comprehensively in the treatment of disabling gastroesophageal reflux requiring gastric bypass after anastomosis.

The strategy under study is objective reflux suppression after fundoplication with the stomach excluded in the following specific context: treatment of disabling gastroesophageal reflux requiring post-bypass surgery in Omega.

The eligible study population will be any adult patient at the investigating center who has undergone one-anastomosis gastric bypass surgery followed by fundoplication of the excluded stomach as part of treatment for disabling post-bypass gastro-oesophageal reflux, resistant to medical treatment and requiring surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patient operated for one anastomosis gastric bypass followed by Fundoplicature with stomach excluded for disabling gastroesophageal reflux requiring surgery within 2 years prior to inclusion;
* Patient in failure of medical treatment;
* Weight loss greater than 50% of excess weight;
* Patient with preoperative objective investigations (gastrojejunal fibroscopy, ph-impedancemetry, abdominal CT scan) of gastroesophageal reflux disease;
* Patient able to understand study-related information and to complete quality-of-life questionnaires in the opinion of the investigator;
* Patient willing to accept study evaluations;
* For women of childbearing age, effective contraception for the duration of the study or negative blood pregnancy test;
* Patient has been informed and has given free, informed and written consent.

Exclusion Criteria:

* Patient with conversion from one anastomosis gastric bypass to Y bypass for disabling gastroesophageal reflux requiring surgery;
* Patient with concomitant hiatal hernia correction for one anastomosis gastric bypass ;
* Patient with secondary one anastomosis gastric bypass ;
* Patient with a deregulated diet;
* Patient under legal protection, or deprived of liberty by judicial or administrative decision;
* Patient unable to understand study information for linguistic, psychological, cognitive or other reasons;
* Women who are or may become pregnant, of childbearing age, without effective contraception or who are breast-feeding;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial that could interfere with the results of the present study;
* Patient not covered by a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate after Fundoplicature with stomach excluded | 2 years
  The primary endpoint is the long-term efficacy of Fundoplicature with stomach excluded in the treatment of disabling Gastroesophageal Reflux Disease requiring Omega post-bypass surgery after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique des Cèdres, Cornebarrieu, France

IPD SHARING:
Plan to Share IPD: No